CLINICAL TRIAL: NCT03531840
Title: Phase II Study of Olaparib in Subjects With Malignant Mesothelioma
Brief Title: Olaparib in People With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180097; 18-C-0097
Record Dates: First submitted 2018-05-18; First posted 2018-05-22 (Actual); Results first posted 2021-03-11 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-03

CONDITIONS: Mesothelioma
Keywords: DNA Mismatch Repair; BAP1; BRCA
MeSH Terms: conditions — Mesothelioma | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Arm 1/Olaparib (Experimental): Twice daily oral olaparib
  Interventions: Drug: Olaparib; Device: ClinOmics

INTERVENTIONS:
Drug: Olaparib — All subjects will take olaparib by mouth twice per day until disease progression or unacceptable toxicity
  Other Names: Lynparza
Device: ClinOmics — Non-significant risk (NSR) device

SUMMARY:
Background:

The drug olaparib may stop cancer cells from fixing damage to their deoxyribonucleic acid (DNA). It has been approved to treat certain cancers in people that were born with a mutation in the breast cancer (BRCA) gene. It has not been approved for treating mesothelioma. But some people with mesothelioma have mutations in a gene, BRCA1 Associated Protein 1 (BAP1) related to BRCA. Researchers want to see if olaparib can work in patients with mutations in this gene. They also want to see if works on mutations in other genes or patients without any mutations. They want to see if olaparib causes mesothelioma tumors to shrink.

Objective:

To study the effect of olaparib on mesothelioma.

Eligibility:

People ages 18 and older with malignant mesothelioma that has already been treated

Design:

Participants will be screened with

Sample of tumor tissue or fluid

Medical history

Physical exam

Blood, heart, and urine tests

Scans and x-rays

Participants will give blood and tissue samples. These will be genetically tested.

The study will be done in 21-day cycles.

Participants will take tables of the study drug 2 times each day. They will get information on what food and drugs to avoid during the study. They will get information about birth control. They will keep a diary of doses and symptoms.

Participants will have blood and urine tests and scans every few weeks.

Participants will be told any important genetic testing results.

Participants will stay in the study until their disease gets worse or the participant or their doctor chooses to stop it.

About 30 days after stopping the study drug, participants will have a follow-up visit. They will have a medical history, physical exam, blood tests, and scans.

Some participants will continue to have scans every 6 weeks.

...

DETAILED DESCRIPTION:
Background:

* Malignant mesothelioma is an invasive and often fatal neoplasm that arises from mesothelium that lines several organs.
* Recent studies have identified germline mutations in the gene encoding breast cancer type 1 (BRCA1) associated protein-1 (BAP1) which can predispose to mesothelioma
* In addition to mesothelioma, germline BAP1 mutations confer increased susceptibility for the development of several other tumors including uveal melanoma, cutaneous melanoma, renal cell cancers and possibly other cancers
* In addition to BAP1, we found several novel germline variants that have previously not been associated with risk of developing mesothelioma.
* As evidenced by recent data derived from ovarian and prostate cancer patients, mutations in deoxyribonucleic acid (DNA) repair genes can define subgroups of cancer patients with distinct vulnerabilities to DNA damage response inhibitors.
* Olaparib is a Poly (ADP-ribose) polymerase (PARP) inhibitor indicated as monotherapy in patients with deleterious or suspected deleterious germline BRCA mutated
* Both established and patient derived mesothelioma cell lines with mutated DNA repair genes are sensitive to olaparib.

Objective:

-Determine the efficacy with respect to objective response rate of olaparib in patients with malignant mesothelioma based on somatic or germline mutation status of DNA repair genes

Eligibility:

* Patients must have progressive, histologically or cytologically confirmed malignant mesothelioma.
* Age greater than or equal to 18 years
* Patients must have received prior platinum and pemetrexed based therapies
* Adequate organ and bone marrow function

Design:

* This is a phase II, single center study of olaparib in subjects with malignant mesothelioma
* All subjects will take olaparib by mouth twice daily until disease progression or intolerable side effects
* Subjects will be assessed for safety (continuously) and efficacy (every 6 weeks)
* Subjects will be analyzed in 3 separate comparison groups according to their mutation status

  * Comparison Group 1: Patients with a germline mutation in DNA repair genes
  * Comparison Group 2: Patients with BAP1 somatic mutations
  * Comparison Group 3: Patients with neither germline mutations nor BAP 1 somatic mutations
* Up to 30 evaluable subjects will be enrolled

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically malignant mesothelioma confirmed by the National Cancer Institute (NCI) Laboratory of Pathology. Patients with pleural, peritoneal, pericardial or tunica vaginalis mesothelioma are eligible.
* Archival tumor samples must be available and sufficient for diagnostic and genetic testing; if archival sample insufficient for testing, subject must have lesions amenable to biopsy and be willing to undergo biopsy.
* Patients must have measurable disease.
* Patients must have progressive disease at study entry
* Patients must have received prior platinum and pemetrexed based therapies. Response to platinum is not an eligibility criterion for enrollment.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of olaparib in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1.
* Patients must have a life expectancy of greater than or equal to 16 weeks
* Patients must have adequate organ and marrow function less than or equal to 5 days prior to Cycle 1 Day 1 (C1D1) as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to greater than or equal to 1,500/mcL without growth factor support
  * platelets greater than or equal to 100,000/mcL
  * hemoglobin greater than or equal to 10 g/dL with no blood transfusion in the past 28 days
  * total bilirubin less than or equal to 1.5 x upper limits of normal (ULN) (unless Gilbert's Disease)
  * Aspartate aminotransferase (AST) Serum glutamic oxaloacetic transaminase (SGOT)/Alanine aminotransferase (ALT) Serum glutamic-pyruvic transaminase (SGPT) less than or equal to 2.5 X institutional upper limit of normal (less than or equal to 5 X ULN in the presence of liver metastases)
  * creatinine clearance greater than or equal to 51 mL/min (calculated using the -Cockcroft-Gault formula.
* Pre-clinical data indicate that olaparib can have adverse effects on embryofetal survival and development. It is further not known whether olaparib or its metabolites are found in seminal fluid. For these reasons:
* Women of childbearing potential and their partners, who are sexually active, must agree to the use of 2 highly effective forms of contraception in combination (male condom plus one other method or must totally/truly abstain from any form of sexual intercourse. This should be started from the signing of the informed consent, throughout their participation in the study and for at least 1 month after the last dose of olaparib.
* Male patients must use a condom during treatment and for 3 months after the last dose of olaparib when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential. Male patients should not donate sperm throughout the period of taking olaparib and for 3 months following the last dose of olaparib.
* Acceptable birth control methods:

  * Total sexual abstinence i.e., refrain from any form of sexual intercourse in line with the patients usual and/or preferred lifestyle. Abstinence must be for the total duration of the study treatment and for at least 1 month (for female patients) or 3 months (for male patients) after the last dose of study treatment. Periodic abstinence (e.g., calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
  * Vasectomised sexual partner PLUS male condom. With participant assurance that partner received post-vasectomy confirmation of azoospermia.
  * Tubal occlusion PLUS male condom
  * Intrauterine Device PLUS male condom. Provided coils are copper-banded.
  * Etonogestrel implants (e.g., Implanon, Norplant) PLUS male condom
  * Normal and low dose combined oral pills PLUS male condom
  * Hormonal shot or injection (e.g., Depo-Provera) PLUS male condom
  * Intrauterine system device (e.g., levonorgestrel-releasing intrauterine system -Mirena) PLUS male condom
  * Norelgestromin/ethinyl estradiol transdermal system PLUS male condom
  * Intravaginal device (e.g., ethinyl estradiol and etonogestrel) PLUS male condom
  * Cerazette (desogestrel) PLUS male condom. Cerazette is currently the only highly efficacious progesterone based pill.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Patients who have received any previous treatment with a Poly (ADP-ribose) polymerase (PARP) inhibitor, including olaparib.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
* Patients with other malignancy documented as occurring within the last 1 year except: adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) documented as curatively treated or under control for greater than or equal to 1 year.
* Patients with features suggestive of Myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML) on peripheral blood smear.
* Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* History of allergic reactions or hypersensitivity attributed to compounds of similar chemical or biologic composition to olaparib or its excipients.
* Patients who have had a whole blood transfusion within 120 days prior to enrollment. (Packed red blood cells and platelet transfusions are acceptable)
* Patients with persistent toxicities (greater than or equal to Common Terminology Criteria for Adverse Events (CTCAE) grade 2) with the exception of alopecia,caused by previous cancer therapy
* Concomitant use of known strong or moderate cytochrome P450, family 3 (CYP3A) inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong CYP3A inducers (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Resting electrocardiogram (ECG) with Fridericia's formula (QTcF) > 470 msec on 2 or more time points within a 24-hour period or family history of long Q wave, T wave (QT) syndrome
* Patients that have had major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Pregnant women are excluded from this study because olaparib has the potential for teratogenic or abortifacient effects. Women must either be post-menopausal or must have a negative pregnancy test (urine or serum) less than or equal to 28 days prior to enrollment and confirmed on day 1 of cycle 1 of study therapy. Postmenopausal is defined as:

Amenorrheic for 1 year or more following cessation of exogenous hormonaltreatments

Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50 years of age

radiation-induced oophorectomy with last menses >1 year ago

chemotherapy-induced menopause with >1-year interval since last menses

surgical sterilisation (bilateral oophorectomy or hysterectomy)

* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib, breastfeeding should be discontinued if the mother is treated with olaparib.
* Immunocompromised patients are excluded.
* Patients who are known to be serologically positive for human immunodeficiency virus (HIV). This includes HIV patients on antiretroviral therapy due to the potential for pharmacokinetic interactions with olaparib.
* Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
* Previous allogeneic hematopoietic stem cell transplant, allogeneic bone marrow transplant or double umbilical cord blood transplant (duCBT)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2020-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2018-C-0097.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data is grouped as specified per protocol.
Groups:
- Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes: Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes
- Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations
- Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations
- Participants Not Classified Under Comparison Groups: Participants With no tumor tissue available for somatic mutation
Period: Overall Study
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations | Participants Not Classified Under Comparison Groups
Started | 5 | 6 | 8 | 4
Completed | 0 | 1 | 3 | 1
Not Completed | 5 | 5 | 5 | 3
Not completed — Death on study | 3 | 2 | 1 | 2
Not completed — Death during follow up | 2 | 3 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Data is grouped as specified per protocol.
Groups:
- Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations; Participants Not Classified Under Comparison Groups: Participants With no tumor tissue available for somatic mutation
- Total: Total of all reporting groups
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations | Participants Not Classified Under Comparison Groups | Total
Number analyzed (Participants) | 5 | 6 | 8 | 4 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 1 | 13
  >=65 years | 1 | 2 | 4 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (14.51) | 61.82 (10.71) | 63.3 (10.5) | 65.3 (4.19) | 61.8 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 0 | 9
  Male | 2 | 3 | 5 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 7 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 5 | 6 | 8 | 4 | 23
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 7 | 3 | 21
  Canada | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Response
Description: Number of participants overall who experienced partial or complete response. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, and the Malignant Pleural Mesothelioma (MPM) criteria. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete Response is disappearance of all target lesions.
Time Frame: 6 months after enrollment of last patient
Population: Data is grouped as specified per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations | Participants Not Classified Under Comparison Groups
Number analyzed (Participants) | 5 | 6 | 8 | 4
Participants
  Partial Response | 1 | 0 | 0 | 0
  Complete Response | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Germline Deoxyribonucleic Acid (DNA) Repair Mutation Who Experienced Partial or Complete Response.
Description: Number of participants with germline deoxyribonucleic acid (DNA) repair mutation who experienced partial or complete response. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, and the Malignant Pleural Mesothelioma (MPM) criteria. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete Response is disappearance of all target lesions.
Time Frame: 6 months after enrollment of last patient
Population: Per protocol, this outcome measure was only assessed in participants in Comparison Group 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes
Number analyzed (Participants) | 5
Participants
  Partial Response | 1
  Complete Response | 0

3. Primary Outcome: Percentage of Participants With Breast Cancer Type 1 Associated Protein-1 (BAP1) Somatic Mutations Who Experienced Partial or Complete Response.
Description: Percentage of participants with germline deoxyribonucleic acid (DNA) repair mutation who experienced partial or complete response. Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, and the Malignant Pleural Mesothelioma (MPM) criteria. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete Response is disappearance of all target lesions.
Time Frame: 6 months after enrollment of last patient
Population: Per protocol, this outcome measure was only assessed in participants in Comparison Group 2.
Measure: Number; unit: percentage of participants
Arm/Group | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations
Number analyzed (Participants) | 6
percentage of participants
  Partial Response | 0
  Complete Response | 0

4. Primary Outcome: Percentage of Subjects With Neither Germline Deoxyribonuclecic Acid (DNA) Repair Mutations Nor Somatic Breast Cancer Type 1 Associated Protein-1 (BAP1) Mutations Who Experienced Partial or Complete Response.
Description: Percentage of subjects with neither germline DNA repair mutations nor somatic BAP1 mutations who experienced partial or complete response.Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, and the Malignant Pleural Mesothelioma (MPM) criteria. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Complete Response is disappearance of all target lesions.
Time Frame: 6 months after enrollment of last patient
Population: Per protocol, this outcome measure was only assessed in participants in Comparison Group 3.
Measure: Number; unit: percentage of participants
Arm/Group | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations
Number analyzed (Participants) | 8
percentage of participants
  Partial Response | 0
  Complete Response | 0

5. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Adverse events were recorded from the study start date until prior to the study completion date, approximately 27 months and 11 days.
Population: Data is grouped as specified per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations: Comparison Group 2 Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations | Participants Not Classified Under Comparison Groups
Number analyzed (Participants) | 5 | 6 | 8 | 4
Participants | 5 | 6 | 8 | 4

6. Secondary Outcome: Number of Participants With Dose Limiting-toxicities (DLT's)
Description: Dose Limiting-toxicities (DLT's) is defined as
Time Frame: 21 days after enrollment of last subject
Population: Data is grouped as specified per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations | Participants Not Classified Under Comparison Groups
Number analyzed (Participants) | 5 | 6 | 8 | 4
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 18 months and 25 days for Group 1, 27 months and 8 days for Group 2, and 26 months and 18 days for both Group 3 and Participants not classified under comparison groups..
Description: Data is grouped as specified per protocol.
Arm/Group | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations | Participants Not Classified Under Comparison Groups
All-Cause Mortality (participants affected / at risk) | 5/5 | 5/6 | 5/8 | 3/4
Serious Adverse Events (participants affected / at risk) | 1/5 | 4/6 | 1/8 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 8/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes (N=5) | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations (N=6) | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations (N=8) | Participants Not Classified Under Comparison Groups (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Eye disorders - Lt orbital solitary (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comparison Group 1:Participants With a Germline Mutation in Deoxyribonucleic Acid (DNA) Repair Genes (N=5) | Comparison Group 2: Participants With BRCA1 Associated Protein-1 (BAP1) Somatic Mutations (N=6) | Comparison Group 3: Participants With Neither Germline Mutations Nor BAP 1 Somatic Mutations (N=8) | Participants Not Classified Under Comparison Groups (N=4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (4) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (10) | 3 (7) | 2 (2) | 2 (7)
Anorexia (Metabolism and nutrition disorders) | 3 (4) | 3 (3) | 4 (4) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 4 (4) | 0 (0)
Creatinine increased (Investigations) | 3 (7) | 2 (5) | 3 (6) | 1 (1)
Dehydration (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (9) | 2 (3) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 1 (1) | 2 (2) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Endocrine disorders - Other, thyrotropin (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, macular degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (5) | 5 (5) | 2 (3) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, cachexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glucosuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3) | 3 (4) | 2 (4) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5) | 2 (2) | 3 (3) | 3 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5) | 5 (9) | 2 (2) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (3)
Keratitis (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (16) | 5 (8) | 6 (17) | 3 (5)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (5) | 6 (7) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (9) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, creatinine clearance decreased (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, skin disorders, others facial erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrush (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 3 (7) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Weight loss (Investigations) | 2 (3) | 1 (2) | 2 (3) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 2 (4) | 0 (0)
Eye disorders - Other, eye disorder, diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, eye disorder, Lt potosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, eye disorder, proptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, vision loss (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders- Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03531840/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03531840/ICF_001.pdf